CLINICAL TRIAL: NCT04809740
Title: Evaluating the Implementation and Impact of Navigator-delivered ePRO Home Symptom Monitoring and Management
Brief Title: Evaluating the Implementation and Impact of Navigator-delivered ePRO System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of South Alabama (Other)
Responsible Party: Principal Investigator, Gabrielle Rocque, Associate Professor of Medicine, Division of Hematology & Oncology; Division of Gerontology, Geriatrics, & Palliative Care, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300007406
Record Dates: First submitted 2020-12-10; First posted 2021-03-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Group (Other): 7,500 Patients from UAB/MCI
  Interventions: Other: Evaluate implementation of navigator-delivered Home ePRO for all cancer patients

INTERVENTIONS:
Other: Evaluate implementation of navigator-delivered Home ePRO for all cancer patients — evaluate implementation of navigator-delivered Home ePRO for all cancer patients across multiple practice sites; 2) examine the barriers, facilitators, and implementation strategies used in implementing navigator-delivered Home ePRO; and 3) assess the impact of Home ePRO on clinical and utilization outcomes

SUMMARY:
1) Evaluate implementation of navigator-delivered Home ePRO for all cancer patients across multiple practice sites; 2) examine the barriers, facilitators, and implementation strategies used in implementing navigator-delivered Home ePRO; and 3) assess the impact of Home ePRO on clinical and utilization outcomes.

DETAILED DESCRIPTION:
Randomized controlled trials by Basch (collaborator) and colleagues demonstrated that weekly electronic home-based PRO symptom monitoring with automated alerts to clinicians (Home ePRO) in cancer patients was associated with reduced healthcare utilization, improved quality of life, and increased overall survival. However, these trials were administered using infrastructure supported by research funding. A knowledge gap remains about optimal implementation strategies for and effectiveness of Home ePROs in real-world settings. To address this gap, investigators from two institutions will conduct a large-scale population-based implementation of an evidence-based Home ePRO intervention for all adult cancer patients receiving chemotherapy, including vulnerable populations such as African Americans, rural residents, and socioeconomically disadvantaged individuals. This implementation will leverage infrastructure from Medicare's payment reform projects (Oncology Care Model, Oncology Care First Model), which require and financially support patient navigators, a natural workforce for Home ePRO implementation. The investigators' hypothesis is that the deployed implementation strategies will result in successful navigator-delivered Home ePRO, which will improve both patient and health system outcomes. Using the Consolidated Framework for Implementation Research (CFIR), this hypothesis will be tested using a hybrid type 2 design with three specific aims: 1) evaluate implementation of navigator-delivered Home ePRO for all cancer patients across multiple practice sites; 2) examine the barriers, facilitators, and implementation strategies used in implementing navigator-delivered Home ePRO; and 3) assess the impact of Home ePRO on clinical and utilization outcomes. In Aim 1, Home ePRO will be evaluated using implementation outcomes (service penetrance, provider adoption/penetration, intervention fidelity). In Aim 2, the investigators will gauge patient and healthcare team perceptions of barriers, facilitators of navigator-led Home ePRO, implementation strategies used to address these barriers, implementation strategy fidelity, and perception of implementation strategy ability to address barriers using an iterative qualitative analysis. In Aim 3, patient-level outcomes (functional status, distress, depression, healthcare utilization, cost, survival) will be evaluated using real-world data sources. The project is innovative because it will be the first study to evaluate real-world implementation of navigator-led Home ePRO for all cancer patients receiving chemotherapy, an approach that is both immediately scalable and sustainable within value-based payment models. The proposed research is significant because it is expected to demonstrate successful implementation of navigator-delivered Home ePRO and effectiveness of the ePRO intervention on diverse patient populations. Furthermore, the project will generate an implementation blueprint of successful implementation strategies that can be easily applied to other patient-reported outcomes, with the potential to positively impact patient care as health care transitions to a value-based system.

ELIGIBILITY:
Inclusion Criteria:

Patient Group:

* Age ≥18
* Cancer patients at participating institution
* Receipt of chemotherapy, targeted therapy, and immunotherapy at participating institution from 2019-2026.

Exclusion Criteria:

- Second opinion only at participating institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Service Penetration | 5 years
  % of eligible patients enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Rocque GB, Dionne-Odom JN, Stover AM, Daniel CL, Azuero A, Huang CS, Ingram SA, Franks JA, Caston NE, Dent AN, Basch EM, Jackson BE, Howell D, Weiner BJ, Pierce JY. Evaluating the implementation and impact of navigator-supported remote symptom monitoring and management: a protocol for a hybrid type 2 clinical trial. BMC Health Serv Res. 2022 Apr 22;22(1):538. doi: 10.1186/s12913-022-07914-6. PMID 35459238